CLINICAL TRIAL: NCT03502863
Title: A Prospective Clinical Study to Evaluate the Effectiveness of Digital Refraction
Brief Title: Clinical Study to Evaluate Effectiveness of Digital Refraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visibly (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPT-1001
Record Dates: First submitted 2018-04-07; First posted 2018-04-19 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Digital refraction (Experimental): Web-based application for obtaining the refractive error and visual acuity of each eye, using a computer and a smart phone
  Interventions: Other: Manual Refraction
- Manual Refraction (Active Comparator): Manual manifest refraction is performed by an eyesore specialist using a phoropter.
  Interventions: Device: Digital refraction

INTERVENTIONS:
Device: Digital refraction — A web-based application for obtaining the refractive error and visual acuity of each eye, using a computer and a smart phone.
  Arms: Manual Refraction
Other: Manual Refraction — Manual refraction and ETDRS chart
  Arms: Digital refraction

SUMMARY:
Prospective, comparative, randomized, non-masked clinical study to compare the a digital refraction with LogMAR VA testing utilizing trial lenses, to standard manual refraction using a Phoropter, and LogMAR VA testing, in accuracy of visual acuity measurement.

DETAILED DESCRIPTION:
A digital refraction tool is a device meant to measure visual acuity and to subjectively measure refractive value for a patient's eye for the conditions of myopia and astigmatism. It is intended for adults aged 22 to 55 years that have no prior correction with up to 3.00 diopters (D) of myopia and up to 2.00 D of astigmatism, or those with prior correction up to 10.00 D of myopia and require an over-refraction of no more than 2.75 D.

LogMAR (ETDRS) chart to measure visual acuity.

The manual manifest refraction is performed by an eyecare specialist using a phoropter.

The LogMAR Visual Acuity chart is used to measure visual acuity. The manual refraction will be used in this study for obtaining the refractive error of each eye.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be between 22 and 55 years of age at the time of consent.
2. Subject must have a refractive error

   1. With no greater than -3.00 D myopia and -2.00 D astigmatism in either eye.
   2. With prior correction of no greater than -10.00 D myopia and requiring over-refraction of no more than 2.75 D in either eye.

5. Subjects with Best Corrected Visual Acuity (BCVA) of 20/32 or better.

Exclusion Criteria:

1. Subjects with diabetes mellitus.
2. Subjects using ophthalmic or systemic corticosteroids.
3. Subjects with autoimmune conditions.
4. Subjects with active corneal or conjunctival infection.
5. Subjects with active corneal, conjunctival, or intraocular inflammation (ie, uveitis).
6. Subjects with diabetic retinopathy.
7. Subjects with glaucoma or ocular hypertension.
8. Subjects with macular degeneration.
9. Subjects with previous ocular surgery.
10. Subjects on antihyperglycemic agents; corticosteroids; hydroxychloroquine (Plaquenil) and chloroquine (Aralen); tamoxifen (Nolvadex).
11. Pregnancy
12. Subjects who, in the judgment of the Investigator, may be inappropriate for the intended study procedures.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
A digital refraction will be compared to standard manual refraction methods (using a phoropter) to the correlation of the two methods. | After the Day 1 Visits
  The difference between testing methods (Manual Refraction with a phoropter versus a digital refraction test) will be analyzed by mean, standard deviation, and 95% confidence interval overall and by the levels of refractive correction (sphere, cylinder, MRSE) and for visual acuity using LogMAR format.

CONTACTS AND LOCATIONS:
Overall Officials: S Lee, Study Director — Sponsor GmbH
Locations (3):
- United States (3):
  - Site 03, Fort Lauderdale, Florida
  - Site 02, Nashville, Tennessee
  - Site 01, Harlingen, Texas